CLINICAL TRIAL: NCT04185181
Title: Virtual Reality Versus Proprioceptive Neuromuscular Facilitation on Postmastectomy Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: doaa atef (Other)
Responsible Party: Sponsor-Investigator, doaa atef, assistant lecturer of physical therapy for surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doaa Atef
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Postmastectomy Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Active Comparator)
  Interventions: Other: virtual reality; Other: complete decogestive therapy
- propreoceptive neuromuscular facilitation (Active Comparator)
  Interventions: Other: proprioceptive neuromuscular facilitation; Other: complete decogestive therapy

INTERVENTIONS:
Other: virtual reality — wii video game based exercise
  Arms: virtual reality
Other: proprioceptive neuromuscular facilitation — PNF with breathing
  Arms: propreoceptive neuromuscular facilitation
Other: complete decogestive therapy — pneumatic compression, manual lymph drainage, skin care and home exercise program

SUMMARY:
This study aimed to compare the therapeutic efficacy of VR and PNF on lymphedema and function in unilateral post-mastectomy lymphedema (UPML) patients. The patients were subdivided into two equal groups, 15 in each. Fifteen patients performed virtual reality-based exercises plus complete decongestive therapy, while the other fifteen patients performed proprioceptive neuromuscular facilitation plus complete decongestive therapy. The volume difference between normal and affected limbs was calculated before and after eight sessions of treatment for both groups by using the circumferential method. And the upper limb function was assessed before and after eight sessions of treatment for both groups by using the Arabic version of the Quick DASH scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients will suffer from unilateral post-mastectomy lymphedema.
* Stage I and stage II lymphedema as defined by the classification of the International Society of Lymphology (The International Society of Lymphology, 2003).
* Patients had no physical therapy before the current treatment or the last time to receive sessions was at least three months ago.

Exclusion Criteria:

* Excluded patients were having musculoskeletal or neurological disorders that would impair performance during training and tests.
* Visual disorders that could affect imitation of video game-based exercise.
* Uncontrolled cardiovascular or pulmonary diseases.
* Psychiatric illness, severe behavior, and cognitive disorders.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
lymphedema volume | 4 weeks
  turncated cone formula using circumferential measurement of both upper limbs
upper limb function | 4 weeks
  quick-disability of arm, shoulder and hand (DASH) scale. minimum score is zero and maximum score is 44. higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: doaa AA abd-el-wahed, A.lecturer, Principal Investigator — assistant lecturer at faculty of physical therapy, Cairo university
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atef D, Elkeblawy MM, El-Sebaie A, Abouelnaga WAI. A quasi-randomized clinical trial: virtual reality versus proprioceptive neuromuscular facilitation for postmastectomy lymphedema. J Egypt Natl Canc Inst. 2020 Jun 15;32(1):29. doi: 10.1186/s43046-020-00041-5. PMID 32537717